CLINICAL TRIAL: NCT02866006
Title: Open-label, Dose-escalation, Multiple Dosing Study to Evaluate the Safety, Tolerability, Immune Response and Pre Efficacy of BVAC-C in Patients With Multiple Metastatic Progressive or Recurrent HPV Type 16 or 18 Positive Cervical Cancer After Failure to Standard Care
Brief Title: Safety and Tolerability Evaluation Study of BVAC-C in Patients With HPV Type 16 or 18 Positive Cervical Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Cellid Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BVAC-C-P1
Record Dates: First submitted 2016-08-09; First posted 2016-08-15 (Estimated); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Uterine Cervical Neoplasms
Keywords: HPV; Type 16, 18; E6E7; Immune therapeutic vaccine
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Topotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- BVAC-C mono(High dose) (Experimental): BVAC-C IV injection at 0, 4, 8th weeks.(HIgh dose)
  Interventions: Drug: BVAC-C
- BVAC-C mono(Intermediate dose) (Experimental): BVAC-C IV injection at 0, 4, 8, 12th weeks.(Half dose)
  Interventions: Drug: BVAC-C
- BVAC-C + Topo Combi (Experimental): BVAC-C IV injection at 0,4,8,12th weeks.(Half dose) Topotecan IV injection at 2, 6, 10, 14th weeks
  Interventions: Drug: BVAC-C; Drug: Topotecan

INTERVENTIONS:
Drug: BVAC-C — Autologous B cells and monocytes transfected with E6E7 gene of HPV
Drug: Topotecan
  Arms: BVAC-C + Topo Combi

SUMMARY:
BVAC-C is an immunotherapeutic vaccine using B-Cell and Monocytes as antigen-presenting cells. This study is consists of 2 parts. Phase I is for safety evaluation, and Phase IIa is for efficacy assessment.

DETAILED DESCRIPTION:
BVAC-C is an immunotherapeutic vaccine using B-Cell and Monocytes as antigen-presenting cells. This study is consists of 2 parts(Phase I, Phase II). Phase I study is Open-label, dose-escalation, multiple dosing study to evaluate the safety, tolerability, immune response and preliminary efficacy of BVAC-C in patients with multiple metastatic progressive or recurrent HPV type 16 or 18 positive cervical cancer after failure to standard care. 9~18 patients will be enrolled In Phase IIa study, which Open-label, sequential assignment multiple dosing study, efficacy, immune response and safety will be evaluated. Total 21 patients will be enrolled in 3 groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients with multiple metastatic progressive or recurrent HPV type 16 or 18 positive cervical cancer
* Patients has received 1 or more platinum based doublet chemotherapy as prior therapy for progressive or recurrent tumor lesion (prior therapy does not include platinum chemotherapy given with radiation therapy for 1st line treatment before progression or recurrence)
* Patients with at least 1 measurable lesion according to RECIST
* Female patients between ages of 20 to 70
* Patients with ECOG performance status between 0 to 2
* Patients meets the blood test standards in the screening test

  * ANC≥1500/μL
  * LLN ≤ALC ≤ULN
  * Platelets≥100,000/μL
  * Hemoglobin> 9g/dL
* Patients meets the blood chemistry test standards in the screening test

  * Serum creatinine ≤ 2.0 mg/dL
  * Calculated creatinine clearance ≥ 50 mL/min
  * Serum bilirubin ≤1.5 x ULN
  * ALT and AST ≤2.5 × ULN (≤ 5 x ULN in patients with liver metastases)
* Patients who has agreed to a medically accepted contraceptive in this clinical trial
* Patients at least three months or more of survival can be expected
* Patients decided to participate in this clinical trial and signed written informed consent

Exclusion Criteria:

* Patients histopathology is a neuroendocrine or small cell carcinoma
* Patients with a history of brain metastasis or signs of brain metastasis
* Patients tested positive in serological tests for hepatitis C virus or hepatitis B virus surface antigen, (HBsAg) or human immunodeficiency virus (HIV)
* Patients with a history of HIV infection
* Patients showing abnormal electrocardiogram , including arrhythmia
* Patients have been administered the drug for other clinical trials within 4weeks before the screening visit
* Patients have been administered any vaccines within 4weeks before the screening visit (eg. hepatitis A, hepatitis B, influenza, Td, etc. )
* Patients have been administered the blood products within 3 months before the screening visit
* Patients have received chemotherapy or radiation therapy within 4weeks before the 1st administration of investigational drug (BVAC-C)
* Patients treated with immunosuppressant or immunomodulatory agents within 6 months before the screening visit
* Patients who have participated in the clinical trial of a therapeutic vaccine or immune therapy within 1 year before the screening visit
* Patients with a history of serious allergic disease or serious side effects of the drug
* Patients who is pregnant or breast-feeding
* Patients researchers has determined that participation in the clinical trial is inappropriate
* Patients suspected to have other primary cancer

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2021-12 (Actual); Study Completion 2022-06 (Actual)

PRIMARY OUTCOMES:
Evaluate DLT with Clinical laboratory tests [Safety] | 12th week from first injection (End of trial)
  Lymphocyte subset, Serum cytokine, NKT/NK cell assay, CD4/CD8 assay
Incidence of Serious Adverse Events assessed with CTCAE [Safety] | 12th week from first injection (End of trial)

SECONDARY OUTCOMES:
Clinical laboratory tests | Screening visit and every 2 weeks from first injection (up to 12th week)
  Blood chemistry, Serology
12-lead ECG | Screening visit and Termination visit (12th week from first injection)
Vital signs | Every 2 weeks from first injection (up to 12th week)
  Blood pressure, Pulse rate, Respiratory rate, Tympanic temperature
Physical examination | Screening, 6th week from first injection, 10th week from first injection and Termination visit (12th week from first injection)
  Body weight

CONTACTS AND LOCATIONS:
Overall Officials: C Y Kang, PH.D, Study Chair — Seoul National University
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Choi CH, Lee JW, Bae DS, Kang ES, Cho D, Kim YM, Kim K, Kim JW, Kim HS, Kim YT, Lee JY, Lim MC, Oh T, Song B, Jeon I, Park M, Kim WH, Kang CY, Kim BG. Efficacy and safety of BVAC-C in HPV type 16- or 18-positive cervical carcinoma who failed 1st platinum-based chemotherapy: a phase I/IIa study. Front Immunol. 2024 Mar 28;15:1371353. doi: 10.3389/fimmu.2024.1371353. eCollection 2024. PMID 38605958